CLINICAL TRIAL: NCT06687044
Title: Sleep Improvement Therapy Affects Pregnancy Outcomes in Chinese Singletons and Twins by Improving Sleep Quality
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Jun Wei (Other)
Responsible Party: Sponsor-Investigator, Jun Wei, Department of Gynecology and Obstetrics, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Sleep improvement therapy
Record Dates: First submitted 2024-11-08; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Gestational Diabetes; Hypertension in Pregnancy; Preterm Labor; NICU Infants
MeSH Terms: conditions — Diabetes, Gestational; Hypertension, Pregnancy-Induced; Obstetric Labor, Premature | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep improvement Therapy group(CBT-I) (Experimental)
  Interventions: Behavioral: Sleep restriction; Behavioral: Stimulation control; Behavioral: Cognitive therapy
- Control group (TAU) (Placebo Comparator)
  Interventions: Behavioral: Sleep principles discussion

INTERVENTIONS:
Behavioral: Sleep restriction — Go to bed before 23pm
  Arms: Sleep improvement Therapy group(CBT-I)
Behavioral: Stimulation control — Avoid drugs, alcohol, caffeine, and nicotine
  Arms: Sleep improvement Therapy group(CBT-I)
Behavioral: Cognitive therapy — Listen to 30 minutes of soothing music every night for 8 weeks
  Arms: Sleep improvement Therapy group(CBT-I)
Behavioral: Sleep principles discussion — The principles of sleep hygiene are discussed, but without the application of stimulus control or sleep restriction
  Arms: Control group (TAU)

SUMMARY:
During pregnancy, the physical and psychological changes of pregnant women, hyperemesis gravidarum, uterine compression, frequent urination, hip or pelvic pain, back pain, leg cramps, gastroesophageal reflux, changes in mental state, and even changes in lifestyle, habits and tastes may affect the sleep of pregnant women. Due to the coexistence of physiological, psychological, social and other complex factors during pregnancy, the incidence of sleep disorders in pregnant women is relatively high, up to 50%, and shows an increasing trend with the increase of gestational week. Not only seriously affect the quality of life of pregnant women, but also may lead to a variety of pregnancy complications, and even lead to adverse pregnancy outcomes. Therefore, early identification, timely diagnosis and treatment of sleep disorders during pregnancy are important measures to improve or even reverse adverse pregnancy outcomes. Although sleep disorders are more common and seriously harmful during pregnancy, people lack of understanding and attention to such diseases, and often regard them as normal clinical manifestations of pregnancy and neglect diagnosis and treatment.

Studies have shown that maternal sleep disorders are associated with hypertensive disorders during pregnancy, preterm birth, and gestational diabetes. Current research objects mainly focus on single pregnancy, twin related research is less.

The purpose of this study is to explore the perinatal sleep health of pregnant women with twin pregnancies, reduce the complications of pregnant women with twin pregnancies and improve the pregnancy outcomes of mothers and infants by improving sleep quality.

ELIGIBILITY:
Inclusion Criteria: (1) Pregnant women aged 18-45 years. (2) Diagnosed with single or twin pregnancy within 12 weeks of pregnancy, report sleep quality problems, agree to participate in the study and sign the informed consent -

Exclusion Criteria:Have a prior serious underlying medical condition (e.g., diabetes, heart disease), mental illness, or other serious sleep disorder

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 300 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Hypertension in pregnancy | From the data of randomization until the date of the end of this pregnancy (up to 50 weeks)
  Pregnancy induced hypertension (PIH) is hypertension that occurs after 20 weeks of gestation in women with previously normal blood pressure.
Gestational diabetes mellitus | From the data of randomization until the date of the end of this pregnancy (up to 50 weeks)
  Gestational diabetes mellitus (GDM) is defined as glucose intolerance of variable degree with onset or first recognition during pregnancy
Preterm labor | From the data of randomization until the date of the end of this pregnancy (up to 50 weeks)
  Preterm labor is parturition that occurs when birth occurs between 28 weeks of gestation and 37 weeks
NICU infants | From the data of randomization until the date of the end of this pregnancy (up to 50 weeks)
  Neonatal NICU occupancy rate

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No